CLINICAL TRIAL: NCT01617655
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of SAR236553/REGN727 in Patients With Heterozygous Familial Hypercholesterolemia and LDL-C Higher or Equal to 160mg/dL With Their Lipid-Modifying Therapy
Brief Title: Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Placebo on Top of Lipid-Modifying Therapy in Patients With Heterozygous Familial Hypercholesterolemia (ODYSSEY HIGH FH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC12732; U1111-1128-5459 (Other: UTN); 2012-001096-37 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Q2W (Placebo Comparator): Placebo for alirocumab subcutaneous (SC) injection every two weeks (Q2W) on top of stable lipid-modifying therapy (LMT) for 78 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Lipid Modifying Therapy (LMT)
- Alirocumab 150 mg Q2W (Experimental): Alirocumab 150 mg SC injection Q2W on top of stable LMT for 78 weeks.
  Interventions: Drug: Alirocumab; Drug: Lipid Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Alirocumab — Solution for subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre filled pen).
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab 150 mg Q2W
Drug: Placebo (for alirocumab) — Solution for subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre filled pen).
  Arms: Placebo Q2W
Drug: Lipid Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9).

Primary Objective of the study:

To evaluate the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels after 24 weeks of treatment in comparison with placebo.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with placebo on LDL-C at other time points
* To evaluate the effects of alirocumab on other lipid parameters
* To evaluate the safety and tolerability of alirocumab

DETAILED DESCRIPTION:
The maximum study duration was planned to be 89 weeks per participant including participants who successfully completed the 78-week treatment period had the possibility to join an open-label extension study (LTS13463, NCT01954394) at the end of the treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with heterozygous familial hypercholesterolemia who were not adequately controlled with their lipid-modifying therapy.

Exclusion criteria:

* Age < 18 years
* LDL-C < 160 mg/dL (< 4.14 mmol/L) at the screening visit (Week-3).
* Fasting serum triglycerides > 400 mg/dL (> 4.52 mmol/L) during the screening period.
* Known history of homozygous familial hypercholesterolemia.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- United States (14):
  - Investigational Site Number 840742, Bell Gardens, California
  - Investigational Site Number 840703, Newport Beach, California
  - Investigational Site Number 840712, Newport Beach, California
  - Investigational Site Number 840743, Northridge, California
  - Investigational Site Number 840734, Washington D.C., District of Columbia
  - Investigational Site Number 840738, Miami, Florida
  - Investigational Site Number 840710, Ponte Vedra, Florida
  - Investigational Site Number 840701, New York, New York
  - Investigational Site Number 840702, Durham, North Carolina
  - Investigational Site Number 840714, Cincinnati, Ohio
  - Investigational Site Number 840705, Philadelphia, Pennsylvania
  - Investigational Site Number 840709, Philadelphia, Pennsylvania
  - Investigational Site Number 840713, Philadelphia, Pennsylvania
  - Investigational Site Number 840736, Dallas, Texas
- Canada (2):
  - Investigational Site Number 124704, Québec
  - Investigational Site Number 124703, Sherbrooke
- Netherlands (5):
  - Investigational Site Number 528713, Amsterdam
  - Investigational Site Number 528701, Amsterdam
  - Investigational Site Number 528704, Groningen
  - Investigational Site Number 528716, Leiden
  - Investigational Site Number 528709, Utrecht
- Russia (9):
  - Investigational Site Number 643706, Arkhangelsk
  - Investigational Site Number 643705, Kazan'
  - Investigational Site Number 643703, Moscow
  - Investigational Site Number 643711, Moscow
  - Investigational Site Number 643708, Moscow
  - Investigational Site Number 643710, Saint Petersburg
  - Investigational Site Number 643709, Saint Petersburg
  - Investigational Site Number 643702, Saint Petersburg
  - Investigational Site Number 643707, Yaroslavl
- South Africa (5):
  - Investigational Site Number 710701, Bloemfontein
  - Investigational Site Number 710704, Bloemfontein
  - Investigational Site Number 710706, Cap Town
  - Investigational Site Number 710702, Parktown
  - Investigational Site Number 710703, Somerset West

REFERENCES:
- [Background] Kastelein JJ, Robinson JG, Farnier M, Krempf M, Langslet G, Lorenzato C, Gipe DA, Baccara-Dinet MT. Efficacy and safety of alirocumab in patients with heterozygous familial hypercholesterolemia not adequately controlled with current lipid-lowering therapy: design and rationale of the ODYSSEY FH studies. Cardiovasc Drugs Ther. 2014 Jun;28(3):281-9. doi: 10.1007/s10557-014-6523-z. PMID 24842558
- [Result] Ginsberg HN, Rader DJ, Raal FJ, Guyton JR, Baccara-Dinet MT, Lorenzato C, Pordy R, Stroes E. Efficacy and Safety of Alirocumab in Patients with Heterozygous Familial Hypercholesterolemia and LDL-C of 160 mg/dl or Higher. Cardiovasc Drugs Ther. 2016 Oct;30(5):473-483. doi: 10.1007/s10557-016-6685-y. PMID 27618825
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Kastelein JJ, Hovingh GK, Langslet G, Baccara-Dinet MT, Gipe DA, Chaudhari U, Zhao J, Minini P, Farnier M. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 monoclonal antibody alirocumab vs placebo in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Jan-Feb;11(1):195-203.e4. doi: 10.1016/j.jacl.2016.12.004. Epub 2016 Dec 28. PMID 28391886
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 centers in 5 countries. A total of 206 participants were screened between June 2012 and May 2013, 99 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction (MI) or ischemic stroke, and intensity of statin treatment. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:2 ratio (placebo:alirocumab) after confirmation of selection criteria. 107 participants were randomized.
Period: Overall Study
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Started | 35 (Randomized) | 72 (Randomized)
Treated | 35 | 72
Completed | 26 | 43
Not Completed | 9 | 29
Not completed — Adverse Event | 2 | 3
Not completed — Poor compliance to protocol | 1 | 4
Not completed — Participants moved | 0 | 4
Not completed — Consent withdrawn by participant | 1 | 1
Not completed — Last visit outside protocol visit window | 1 | 10
Not completed — Site closure | 3 | 5
Not completed — Other than specified above | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo Q2W: Placebo for alirocumab SC injection Q2W on top of stable LMT for 78 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W | Total
Number analyzed (Participants) | 35 | 72 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.2) | 49.8 (14.2) | 50.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 37 | 50
  Male | 22 | 35 | 57
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  mg/dL | 201 (43.4) | 196.3 (57.9) | 197.8 (53.4)
Calculated low density lipoprotein cholesterol (LDL-C) in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 5.205 (1.125) | 5.083 (1.499) | 5.123 (1.382)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - ITT Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off- treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.6 (4.9) | -45.7 (3.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -39.1, 95% CI 2-sided [-51.1 to -27.1] — Alirocumab vs Placebo

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.6 (5) | -45.5 (3.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -38.9, 95% CI 2-sided [-51 to -26.9] — Alirocumab vs Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.6 (4.6) | -46.9 (3.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -40.3, 95% CI 2-sided [-51.4 to -29.3] — Alirocumab vs Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.6 (4.6) | -46.9 (3.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -40.3, 95% CI 2-sided [-51.4 to -29.2] — Alirocumab vs Placebo

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 34 | 69
percent change | -8.7 (3.8) | -39 (2.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -30.3, 95% CI 2-sided [-39.7 to -20.9] — Alirocumab vs Placebo

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 34 | 69
percent change | -8.7 (3.9) | -38.9 (2.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -30.2, 95% CI 2-sided [-39.7 to -20.7] — Alirocumab vs Placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.2 (4.3) | -41.9 (3.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -35.8, 95% CI 2-sided [-46.3 to -25.3] — Alirocumab vs Placebo

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.1 (4.3) | -41.7 (3.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -35.5, 95% CI 2-sided [-46.2 to -24.9] — Alirocumab vs Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline total-C value on- or off-treatment (total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -4.8 (3.6) | -33.2 (2.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -28.4, 95% CI 2-sided [-37.3 to -19.6] — Alirocumab vs Placebo

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 34 | 69
percent change | -9 (3.7) | -39.2 (2.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -30.2, 95% CI 2-sided [-39.2 to -21.1] — Alirocumab vs Placebo

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -6.9 (4.3) | -41.4 (3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -34.5, 95% CI 2-sided [-44.8 to -24.1] — Alirocumab vs Placebo

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -5.2 (3.5) | -33 (2.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -27.8, 95% CI 2-sided [-36.2 to -19.4] — Alirocumab vs Placebo

13. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including all available post-baseline data from week 4 to week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -3 (5.9) | -42.1 (4.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -39.1, 95% CI 2-sided [-53.6 to -24.6] — Alirocumab vs Placebo

14. Secondary Outcome: Percentage of Very High Cardiovascular (CV) Risk Participants Achieving Calculated LDL-C < 70 mg/dL (<1.81 mmol/L) or High CV Risk Participants Achieving Calculated LDL-C < 100 mg/dL (<2.59 mmol/L) at Week 24 - ITT Analysis
Description: Very high CV risk participants: Heterozygous Familial Hypercholesterolemia (heFH) participants with coronary heart disease (CHD) or CHD risk equivalents. High CV risk participants: heFH participants without CHD or CHD risk equivalents. CHD risk equivalent: peripheral arterial disease, ischemic stroke, moderate chronic kidney disease (estimated glomerular filtration rate, 30 to <60 ml/minute/1.73 m^2 of body-surface area), or diabetes mellitus plus 2 or more additional risk factors (hypertension; ankle-brachial index of ≤0.90; microalbuminuria, macroalbuminuria, or a urinary dipstick result of >2+ protein; preproliferative or proliferative retinopathy or laser treatment for retinopathy; or a family history of premature CHD). Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percentage of participants | 5.7 | 41.0
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0016, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 11.7, 95% CI 2-sided [2.5 to 53.5] — Alirocumab vs Placebo

15. Secondary Outcome: Percentage of Very High CV Risk Participants Achieving Calculated LDL-C < 70 mg/dL (<1.81 mmol/L) or High CV Risk Participants Achieving Calculated LDL-C < 100 mg/dL (<2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percentage of participants | 5.7 | 41.4
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0014, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 11.9, 95% CI 2-sided [2.6 to 54.9] — Alirocumab vs Placebo

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -8.7 (5) | -23.5 (3.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0164, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -14.8, 95% CI 2-sided [-26.9 to -2.7] — Alirocumab vs Placebo

17. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on-or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | 3.9 (2.7) | 7.5 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2745, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = 3.7, 95% CI 2-sided [-2.9 to 10.2] — Alirocumab vs Placebo

18. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -1.9 (4.8) | -10.5 (3.3)

19. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24 - ITT Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on-or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 34 | 69
percent change | 2 (2.1) | 5.6 (1.5)

20. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -1.5 (5.1) | -23.2 (3.6)

21. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | 8.0 (3.4) | 7.9 (2.4)

22. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 20
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -4.4 (5.1) | -9.4 (3.7)

23. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 34 | 69
percent change | 1.1 (2.2) | 4.6 (1.5)

24. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percentage of participants | 2.9 | 32.4

25. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percentage of participants | 2.9 | 32.6

26. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -2.9 (6.1) | -42.0 (4.4)

27. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM model including all available post-baseline data from Week 4 to Week 78 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 78
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo Q2W: Participants exposed to placebo Q2W on top of stable LMT (mean exposure of 78 weeks).
- Alirocumab 150 Q2W: Participants exposed to Alirocumab 150 mg Q2W on top of stable LMT (mean exposure of 78 weeks).
Arm/Group | Placebo Q2W | Alirocumab 150 Q2W
Number analyzed (Participants) | 35 | 71
percent change | 1.2 (6.4) | -37.9 (4.5)

28. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 78 i.e. up to 21 days after last injection.
Time Frame: From Baseline to Week 78
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 35 | 71
percent change | -0.2 (6.2) | -40.9 (4.5)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit in the study regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent that is AEs that developed/worsened during the 'treatment-emergent period' (from the first double-blind injection up to the day of the last injection + 70 days or up to first intake in the extension study, whichever came first).
Groups:
- Placebo Q2W: Participants exposed to placebo Q2W on top of stable LMT (mean exposure of 71 weeks).
- Alirocumab 150 Q2W: Participants exposed to Alirocumab 150 mg Q2W on top of stable LMT (mean exposure of 68 weeks).
Arm/Group | Placebo Q2W | Alirocumab 150 Q2W
Serious Adverse Events (participants affected / at risk) | 4/35 | 10/72
Other Adverse Events (participants affected / at risk) | 20/35 | 39/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=35) | Alirocumab 150 Q2W (N=72)
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=35) | Alirocumab 150 Q2W (N=72)
Nasopharyngitis (Infections and infestations) | 4 | 10
Influenza (Infections and infestations) | 1 | 9
Bronchitis (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 5
Sinusitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 5
Headache (Nervous system disorders) | 0 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Injection site reaction (General disorders) | 2 | 6
Fatigue (General disorders) | 0 | 5
Blood uric acid increased (Investigations) | 2 | 0

LIMITATIONS AND CAVEATS:
Manual reclassification was done by the Sponsor for the "other reasons" of non-completion of study as specified in the electronic case report form (eCRF).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.